CLINICAL TRIAL: NCT06743464
Title: Effect of Perioperative Oral Rifaximin on Early Graft Dysfunction in Adult Living Donor Liver Transplant: An Open Label Randomized Control Trial
Brief Title: Effect of Perioperative Oral Rifaximin on Early Graft Dysfunction in Adult Living Donor Liver Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-LDLT-03
Record Dates: First submitted 2024-11-25; First posted 2024-12-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-11

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin+SOC (Experimental): Preoperative Rifaximin supplementation 550 mg twice daily from preoperatively 2 weeks to post op POD 1 to 7 SOC (Standard of care) means both group will recieve similar post of care which is standard protocol at ILBS.
  Interventions: Drug: Rifaximin 550 MG; Other: SOC
- Non Rifaximin + SOC (Active Comparator): SOC (Standard of care) means both group will recieve similar post of care which is standard protocol at ILBS.
  Interventions: Other: SOC

INTERVENTIONS:
Drug: Rifaximin 550 MG — Preoperative Rifaximin supplementation 550 mg twice daily from preoperatively 2 weeks to post op POD 1 to 7
  Arms: Rifaximin+SOC
Other: SOC — SOC means Standard of care which means that the patient will revieve standard post op care followed at our insitute and other hospitals in India.

SUMMARY:
Liver transplantation has been a lifesaving treatment for individuals with end stage liver disease and acute liver failure. However, initial poor function of a liver allograft after liver transplantation, termed early graft dysfunction (EGD), has been associated with increased allograft loss or mortality after transplantation. EGD in LDLT is multifactorial. Factors affecting EGD are GRWR, ischemia reperfusion injury, recipient metabolic demand, graft quality, graft inflow and outflow. Studies shows that the incidence of EGD is 15-38%. It is associated with increased allograft loss & mortality. Rifaximin is an antibiotic that reduces EGD by 50% as shown by 2 studies but this study was done in DDLT setting and rifaximin was given in the pretransplant group.

In this investigators will study the effect of perioperative oral rifaximin on early graft dysfunction in adult living donor liver transplant.

DETAILED DESCRIPTION:
Methodology:

* Study population: All patients undergoing adult living donor liver transplant recipients
* Study design: Open label Randomized control Study
* Study period: After ethical board clearance, all LDLT recipients satisfying inclusion criteria till June 2025
* Sample size: n=100

  * Intervention: Preoperative Rifaximin supplementation 550 mg twice daily from preoperatively 2 weeks to post op POD 1 to 7
  * Monitoring and assessment: Not valid
  * Adverse effects: No adverse effect is expected to occur out of study protocols. except vomiting, headache, dizziness, nausea
  * Stopping rule Not valid (b) Expected outcome of the project: Perioperative oral rifaximin decreases early allograft dysfunction in recipients of adult living donor liver transplant. (c) Ethical issues in the study and plans to address these issues: None expected

ELIGIBILITY:
Inclusion Criteria:

* All recipients (adults) undergoing living donor liver transplant in ILBS.

Exclusion Criteria:

* Negative consent

  * Hypersensitivity to Rifaximin
  * Patients undergoing retransplant
  * ALF, ACLF
  * Pediatrics patients
  * Patients on rifaximin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative oral rifaximin on early graft dysfunction in adult living donor liver transplant. | 9 months
  The study aims to see the effect of peri-operative (before transplant and post transplant) rifaximin on early graft dysfunction. Preoperatively investigators will be giving Tab rifaximin supplementation 550 mg twice daily from preoperatively 2 weeks to post op POD 1 to 7 while the other arm will not be given rifaximin.
  Early graft dysfunction is identified using modified altoff criteria, Pamecha et al. creteria(Early graft dysfunction in diseased donor liver transplant and living donor liver transplant)
  1. T. Bilirubin >10
  2. Urea
  3. INR > 1.6
  4. AST/ALT > 2000

SECONDARY OUTCOMES:
To evaluate the effect of rifaximin on early graft dysfunction | 9 months
  Investigators will study the indirect markers for early graft dysfuntion which were recently discovered and the role of rifaximin on the markers. Investigators will do all this in the living donor liver transplant setting
Ischemia reperfusion injury markers (Cathepsin G, CD 86) | 9 months
  Investigators will study the indirect markers for early graft dysfuntion which were recently discovered and the role of rifaximin on the markers. Investigators will do all this in the living donor liver transplant setting
EAD (IL6, IL17) | 9 months
  Investigators will study the indirect markers for early graft dysfuntion which were recently discovered and the role of rifaximin on the markers. Investigators will do all this in the living donor liver transplant setting
To study the effect of perioperative oral rifaximin on infectious complications, EGD related graft loss and in-hospital mortality. | 9 months
  Investigators will study the indirect markers for early graft dysfuntion which were recently discovered and the role of rifaximin on the markers. Investigators will do all this in the living donor liver transplant setting

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India